CLINICAL TRIAL: NCT05661877
Title: Effectiveness of an Online Education Material to Improve Dengue Knowledge and Health-Seeking Intention Among the General Population: An Online Randomized Controlled Trial Via Facebook
Brief Title: Effectiveness of a Online Education Material to Improve Dengue Knowledge and Health-Seeking Intention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2022104-11592
Record Dates: First submitted 2022-11-14; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Dengue
Keywords: dengue; gamification; mobile application; knowledge; health-seeking
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DengueAid intervention group (Experimental): The participants in this arm would be given the DengueAid mobile app which can be downloaded through Google Play
  Interventions: Other: DengueAid mobile application
- MyHealth website control group (Active Comparator): The participants in this arm would be required to use the MyHealth dengue website
  Interventions: Other: MyHealth website

INTERVENTIONS:
Other: DengueAid mobile application — •Education materials regarding dengue fever and self-care. The education section (My Dengue Knowledge) consists of seven modules (dengue essentials, risk, symptoms, aedes mosquito, self-care, prevention and interesting facts) with gamification properties. Each module contains a series of multiple-choice questions. After answering each question, the user would be instantly notified if they had answered the question correctly and be provided with some facts related to the question. A progress meter would allow users to keep track of each module answered. A medal would be awarded to users who have completed 100% of each module. The self-care section consists of basic information about dengue fever and points to look out for self-care. It contains information on dengue fever phases, signs of dengue, importance of keeping hydrated, complementary therapy, medicine to avoid and prevention practices.
  Arms: DengueAid intervention group
Other: MyHealth website — MyHealth is developed by Ministry of Health, Malaysia (http://www.myhealth.gov.my/en/dengue-fever/) to provide information on dengue.
  Arms: MyHealth website control group

SUMMARY:
Dengue is an endemic infectious disease in Malaysia. Delays in seeking treatment and improper self-care contribute to dengue complications and mortality. A mobile app (Dengue Aid) was developed to educate and empower patients to perform evidence-based self-care when having dengue fever. DengueAid is hypothesised to improve people's knowledge and health-seeking intention on dengue. This will be evaluated via an online randomised controlled trial. Adults aged 18 and above who have Facebook, an android smartphone and understand either English or Malay language will be recruited through Facebook advertisements. Eligible participants would be randomized to either using the DengueAid app (intervention) or MyHEALTH website (control). An online randomizer tool will be used to randomize participants into the intervention or control group. Participants in both arms would complete a post-intervention online questionnaire (knowledge and health-seeking intention) three days after recruitment.

DETAILED DESCRIPTION:
The public have shown increasing interest in having health information disseminated to them through smartphones. The current usage of health-related smartphone apps was over 500 million people. In addition, studies have shown that the use of gamification produced positive effect on users' engagement in learning about health and led to positive change in the behaviour for their health and wellness. Several previous studies have shown the effectiveness of mobile applications in promoting health related information. A pilot randomized control trial among coronary heart disease (CHD) patients found that participants in the intervention group (Care4Heart app) showed better overall CHD knowledge levels than participants in the control group (website of Singapore Heart Foundation).

For dengue fever, an integrated mobile health app (Mozzify) was developed and may improve knowledge on dengue fever and promote dissemination and sharing of information on dengue fever among the public and health practitioners. During the development, suggestions to improve the engagement of the app included the addition of games to encourage the public to use it more frequently. Adding to this, the concept of gamification is increasingly being used in health education applications since 2010. Studies have shown that the use of gamification produced positive effect on users' engagement in learning about health and led to positive change in the behaviour for their health and wellness.

As both mobile applications and gamification show increasing importance in the field of mHealth, the DengueAid app was developed to improving monitoring of the disease and knowledge on dengue fever. Previous studies on the effectiveness of a gamified mobile app to improve dengue knowledge was limited to none. In this era of digitalization, an effective gamified mobile intervention for dengue fever which consistently affect the Malaysian population should be developed. Hence, for this study, the effectiveness of DengueAid in improving dengue knowledge among the public will be evaluated through a randomized control trial (RCT).

The sample size was decided on based on previous literature involving the use of a gamified mobile application to improve knowledge on oral health. For a full RCT, using mean and standard deviation values from a previous study (Control Group 13.1 ± 1.6, Intervention Group 14.3 ± 2.0) with 90% power and alpha of 0.05, the estimated sample size is 48 in each arm. Considering a 20% dropout rate the final number of participants recruited would be 116 (58 in each arm).

The study will be advertised on a social media platform (Facebook). Lay public who are interested to join the study will click on a link in the advertisement. The participants will then read the study information sheet and undergo an eligibility check to determine if they are suitable to join the study. Participants who have hearing and speech impairment, cognitive impairment, had dengue before and healthcare staff would be excluded from the study. Participants who are eligible would then have to complete a consent form and provide sociodemographic details. They will then be randomized using an online randomizer to either intervention or control groups. They will be given three days to complete using the intervention/control materials.

Participants in both study arms, would be given three days to complete the online education material (intervention: DengueAid app; control: MyHEALTH website). The research assistant will send an online questionnaire three days after the enrollment day. The questionnaire consists of questions on knowledge on dengue fever based on the modules and content of the DengueAid app as well as questions on health-seeking intention. The questionnaire will be developed using REDCap. Each participant will be compensated with RM30 once they completed the post-intervention online questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Have a social media account
* Have an android smartphone
* Understand English or Malay

Exclusion Criteria:

* Hearing and speech impairment
* Cognitive impairment
* Had dengue before
* Healthcare staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-05-06 (Estimated); Study Completion 2023-05-06 (Estimated)

PRIMARY OUTCOMES:
Knowledge on Dengue | 3 days follow up after enrollment
  Mean knowledge score on dengue (0 to 25, higher score means better outcome)

SECONDARY OUTCOMES:
Health-seeking intention when having dengue fever | 3 days follow up after enrollment
  1. First doctor's visit (medical attention)
     - Percentage of participant agreed to the question "I will see a doctor when I have fever and if there are dengue cases in my neighbourhood."
  2. Follow-up doctors visit (medical attention)
     - Percentage of participant agreed to the question "I will follow doctor's advice and attend all follow ups when diagnosed with dengue"
  3. Emergency doctors visit due to warning signs (medical attention)
     - Percentage of participant agreed to the question "I will seek medical attention immediately if I have either one of the warning signs of dengue such as abdominal pain, blood in stool/vomit, bleeding gums/nose, persistent vomiting/diarrhoea, drowsiness or irritability."
  4. Complementary and alternative medicine (self-care)
     - Percentage of participant agreed to the question on CAM
  5. Medicine and supplements (self-care) - Percentage of participant agreed to the question on medicine and supplements

CONTACTS AND LOCATIONS:
Overall Officials: Chin Hai Teo, Principal Investigator — Universiti Malaya
Locations (1):
- University of Malaya Medical Centre, Kuala Lumpur, Malaysia